CLINICAL TRIAL: NCT06110065
Title: CT-guided Pudendal Nerve Cryoneurolysis for Palliation of Malignancy-induced Pelvic Pain
Status: Not yet recruiting | Type: Observational
Sponsor: University of Arizona (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00002955
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Malignancy-induced Pelvic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort 1
  Interventions: Drug: CT-guided Pudendal Nerve Cryoneurolysis; Drug: Percutaneous image-guided cryoneurolysis

INTERVENTIONS:
Drug: CT-guided Pudendal Nerve Cryoneurolysis — CT-guided bilateral pudendal nerve cryoneurolysis involves using advanced imaging technology to precisely target and freeze the pudendal nerves, which are responsible for transmitting pain signals.
Drug: Percutaneous image-guided cryoneurolysis — Percutaneous image-guided cryoneurolysis focuses on using extremely cold temperatures to alleviate pain originating from the pudendal nerves. This method has demonstrated extended pain relief compared to alternatives like injections or catheters. Additionally, it presents a lower risk of certain complications.

SUMMARY:
We want to study if a new treatment called "CT-guided bilateral pudendal nerve cryoneurolysis" can help people with severe and long-lasting pain in the pelvic area caused by cancer. We will closely follow and observe patients who undergo this treatment to see if it works well, what results it gives, and if there are any problems or side effects. "Percutaneous image-guided cryoneurolysis" involves using very cold temperatures to treat the nerves causing the pain. This method has been found to provide longer pain relief compared to injections or catheters, and it also has a lower risk of certain complications.

We are conducting a study to assess the effectiveness of two different treatments for severe and persistent pelvic pain caused by cancer. The first treatment, known as "CT-guided bilateral pudendal nerve cryoneurolysis," involves using advanced imaging technology to precisely target and freeze the pudendal nerves, which are responsible for transmitting pain signals. By closely monitoring patients who receive this treatment, we aim to evaluate its efficacy, outcomes, and potential side effects.

On the other hand, the second treatment approach, referred to as "Percutaneous image-guided cryoneurolysis," focuses on using extremely cold temperatures to alleviate pain originating from the pudendal nerves. This method has demonstrated extended pain relief compared to alternatives like injections or catheters. Additionally, it presents a lower risk of certain complications. Through our study, we seek to gain insights into the effectiveness and safety of both treatment methods, enhancing our understanding of how to address the challenging issue of cancer-related pelvic pain.

The study will enroll patients who are dealing with severe and persistent pelvic pain from cancer. All patients will undergo the CT-guided bilateral pudendal nerve cryoneurolysis first type of treatment and if it is not effective in relieving the pain, they will be offered to undergo the second treatment called Percutaneous image-guided cryoneurolysis.

Both of these treatments are done as standard of care. This research study will not alter standard of care. Subjects will only be enrolled into this study if they are already undergoing CT-guided bilateral pudendal nerve cryoneurolysis followed up with Percutaneous image-guided cryoneurolysis, as needed. This is a prospective study of these two treatments following patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

Those already scheduled for a CT-guided bilateral pudendal nerve cryoneurolysis as standard of care Age ≥18 years old Active or history of pelvic cancer malignancy Poor pelvic pain control with current therapy (pain from cancer malignancy) Pain in distribution of the pudendal (genital) nerves from cancer malignancy

Exclusion Criteria:

Pain in distribution of the pudendal nerves from nonmalignant etiology Patients with pain from other medical conditions besides cancer/cancer malignancy will not be included (cancer-related pain from cancer malignancy in the genital region is considered).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Interventional Radiology Oncology clinic
Sampling Method: Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Improvement | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Shamar J Young, MD, Principal Investigator — University of Arizona - Department of Medical Imaging
Locations (1):
- University of Arizona, Tucson, Arizona, United States